CLINICAL TRIAL: NCT02247492
Title: BIOTRONIK - SaFety and Performance Registry for an All-comers Patient Population With the Limus Eluting Orsiro Stent System Within Daily Clinical Practice - III and Vulnerable Inflammation Parameter Registry
Brief Title: BIOFLOW-III VIP Russia Registry Orsiro Stent System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Biotronik Russia (Industry)
Responsible Party: Sponsor
Other Study IDs: G1406
Record Dates: First submitted 2014-09-17; First posted 2014-09-25 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Coronary Artery Diseases
Keywords: International; Multicenter; Observational registry; Orsiro Drug Eluting Stent (DES); Stenting; Treatment of coronary artery disease; Coronary revascularization; Percutaneous Coronary Intervention (PCI); STEMI; NSTEMI; Ischemia; Angina; Acute Myocardial Infarction (AMI); Small Vessels; Chronic Total Occlusion (CTO
MeSH Terms: conditions — Coronary Artery Disease; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Ischemia; Angina Pectoris

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Orsiro

SUMMARY:
Clinical evaluation of the Orsiro LESS in subjects requiring coronary revascularization with Drug Eluting Stents (DES). Along with it, an explanatory (hypothesis-finding) problem will be investigated, whether the patient's body inflammation status correlates with the clinical outcome.

DETAILED DESCRIPTION:
For the majority of Coronary Artery Disease (CAD) treatment with Percutaneous Transluminal Coronary Angioplasty (PTCA) provides high initial procedure success. However, the medium to long-term complications range from rather immediate elastic coil or vessel contraction to longer processes like smooth muscle cell proliferation and excessive production of extra cellular matrix, thrombus formation and atherosclerotic changes like restenosis or angiographic re-narrowing. The reported incidence of restenosis after PTCA ranges from 30 to 50%. Such rates of recurrence have serious economic consequences. Bare Metal Stents (BMS), designed to address the limitations of PTCA, reduced the angiographic and clinical restenosis rates in De Novo lesions compared to PTCA alone and decreased the need for CABG. BMS substantially reduced the incidence of abrupt artery closure, but restenosis still occurred in about 20 to 40% of cases, necessitating repeat procedures.

The invention of Drug Eluting Stents (DES) significantly improved on the principle of BMS by adding an antiproliferative drug (directly immobilized on the stent surface or released from a polymer matrix), which inhibits neointimal hyperplasia. The introduction of DES greatly reduced the incidence of restenosis and resulted in better safety profile as compared to BMS with systemic drug administration. These advantages and a lower cost compared to surgical interventions has made DES an attractive option to treat coronary artery disease.

Therefore this observational registry has been designed for the clinical evaluation of the ORSIRO LESS requiring coronary revascularization with DES. It is designed to investigate and collect clinical evidence for the clinical performance and safety of the Orsiro Drug Eluting Stent System in an all-comers patient population in daily clinical practice.

Along with it, an explanatory (hypothesis-finding) problem will be investigated, whether the patient's body inflammation status correlates with the clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic coronary artery disease
* Subject signed informed consent for data release
* Subject is geographically stable and willing to participate at all follow up assessments
* Subject is ≥ 18 years of age

Exclusion Criteria:

* Subject did not sign informed consent
* Pregnancy
* Known intolerance to aspirin, clopidogrel, Ticlopidine, heparin or any other anticoagulant/antiplatelet therapy required for PCI, stainless steel, Sirolimus or contrast media
* Planned surgery within 6 months after PCI unless dual antiplatelet therapy will be maintained
* Currently participating in another study and primary endpoint not reached yet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects requiring coronary revascularization with Drug Eluting Stents (DES)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-04-14 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | 12 months
  Composite of cardiac death, target vessel Q-wave or non Q-wave Myocardial Infarction (MI), Coronary Artery Bypass Graft (CABG) and clinically driven Target Lesion Revascularization (TLR).

SECONDARY OUTCOMES:
Target Lesion Failure (TLF) | 6 and 36 months
  Composite of cardiac death, target vessel Q-wave or non-Q wave Myocardial Infarction (MI), Emergent Coronary Artery Bypass Graft (CABG), clinically driven Target Lesion Revascularization (TLR)
Target Vessel Revascularization (TVR) | 6 and 36 months
  Any repeat revascularization of the target vessel.
Target Lesion Revascularization (TLR) | 6 and 36 months
  Defined as any repeat revascularization of the target lesion.
Stent Thrombosis | 6, 12 and 36 months
  Definite, Probable and Possible Stent Thrombosis
Clinical Device Success | participants will be followed for the duration of hospital stay, an expected average of 1 day
  Successful delivery and deployment of the investigational stent (s) at the intended target lesion and successful withdrawal of the stent delivery system with attainment of a final residual stenosis of less than 50% by visual estimation and without use of device outside the assigned treatment strategy.
Clinical procedural success | up to seven days
  Successful delivery and deployment of the investigational stent (s) at the intended target lesion and successful withdrawal of the stent delivery system with attainment of a final residual stenosis of less than 50% by visual estimation and without using any adjunctive device without the occurrence of ischemia-driven major adverse cardiac event during the hospital stay to a maximum of the first seven days post index procedure.
  In case of multiple lesions treatment, all treated lesions must meet the clinical procedural success.
Vulnerable Inflammation Parameter (VIP) | up to 36 months
  VIP registered ad Endotoxin concentration in patients blood serum

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny Kretov, Dr., Principal Investigator — Novosibirsk Research Institute for Circulation
Locations (7):
- Russia (7):
  - Research Institute for Complex Problems of Cardiovascular Diseases, Kemerovo
  - Regional Clinical Hospital, Nizhny Novgorod
  - Novosibirsk Scientific Research Institute of Circulation Pathology, Novosibirsk
  - City Emergency Clinical Hospital of Rostov-on-Don, Rostov-on-Don
  - North-West Federal Medical Research Center named after V.A. Almazov, Saint Petersburg
  - Institute of Cardiology, Tomsk Medical Research, Tomsk
  - Ural Institute of Cardiology, Yekaterinburg